CLINICAL TRIAL: NCT04267822
Title: Randomized, Double-blind, Placebo-controlled Trial of the Safety, Tolerability, and Efficacy of RV521 in the Treatment of Adult Subjects Who Have Undergone Hematopoietic Cell Transplantation (HCT) With a Documented Upper Respiratory Tract Infection (URTI) With Respiratory Syncytial Virus (RSV)
Brief Title: Study of RV521 in the Treatment of Adult Subjects Who Have Undergone HCT With an URTI With RSV
Acronym: REVIRAL2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REVC006; C5241011 (Other: Pfizer)
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: RSV Infection; Stem Cell Transplant Complications; Lower Resp Tract Infection
Keywords: RV521; lower respiratory tract complication; HCT; hematopoietic cell transplantation; LRTI; Respiratory tract infection; immunocompromise
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Respiratory Tract Infections | interventions — sisunatovir

STUDY DESIGN:
Intervention Model Description: A Phase 2, international, multicenter, randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigators, Sponsor, Independent Adjudication Committee members, and any personnel involved in the subject's care, assessment, monitoring, data collection, or analysis will be blinded to the subject treatment assignment throughout the conduct of the study. Exceptions to this are limited to a fire-walled-protected, unblinded Data Safety Monitoring Board (DSMB) statistician at the Contract Research Organization (CRO) who will prepare output for the closed session of all DSMB meetings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RV521 Capsules (Experimental): RV521 is formulated as a dry powder blend of RV521 drug substance with mannitol as excipient. They are a white, opaque capsule and administered orally.
  Interventions: Drug: RV521 oral tablet
- RV521 Placebo Capsules (Placebo Comparator): RV521 placebo capsules will contain mannitol and microcrystalline cellulose only. They are a white, opaque capsule and administered orally.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: RV521 oral tablet — Each RV521 dose is four 50 mg dry powder blend capsules, taken orally twice daily for 10 days (20 doses total; 80 capsules total)
  Other Names: sisunatovir
  Arms: RV521 Capsules
Drug: Placebo oral tablet — Each placebo dose is four capsules, taken orally twice daily for 10 days (20 doses total; 80 capsules total)
  Other Names: vehicle
  Arms: RV521 Placebo Capsules

SUMMARY:
RV521 is to being developed to treat RSV infection and disease in susceptible individuals at high risk for complications. This is an international, multicenter, placebo-controlled study. Eligible subjects are adults with a documented symptomatic RSV infection who have undergone HCT transplantation and are moderately to severely immunocompromised. Qualified subjects will be randomized in a 1:1 ratio to receive RV521 or placebo, twice daily for 10 days.

DETAILED DESCRIPTION:
The purpose of this study is to compare the viral load, safety, tolerability, and clinical efficacy of RV521 compared to placebo. This is a Phase 2, international, multicenter, randomized, double-blind, placebo-controlled study. Up to 200 adult subjects with a documented symptomatic RSV URTI who have undergone HCT within 1 year of randomization and who are moderately to severely immunocompromised will be randomized.

Qualified subjects will be randomized in a 1:1 ratio to receive RV521 capsules or matching placebo twice daily for 10 days. After the completion of the 10-day double-blind treatment period, subjects will be followed for an additional 28 days. Study drug may be taken on an outpatient or inpatient basis, depending on clinical status and site practices. Randomization will be stratified by type of HCT graft and ALC count. There are 9 clinic visits planned for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Has undergone autologous or allogeneic HCT using any conditioning regimen within 1 year of randomization. Subjects who have undergone HCT more than 1 year before Randomization are eligible if all other inclusion/exclusion criteria are satisfied and under at least one of the following conditions:

   1. Diagnosed with Chronic Graft-vs-Host Disease (GVHD), or
   2. Has used systemic corticosteroids in the 30 days prior to RSV infection
2. Has moderate to severe immunocompromise, defined as a score ≥ 5 on the ISI-RSV and/or an ALC of ≤ 500 cells/ mm3
3. Documentation of positive RSV infection in the upper airway

Exclusion Criteria:

1. Use of non-marketed investigational agents within 30 days, OR use of an investigational monoclonal anti-RSV antibodies within 4 months or 5 half-lives of screening, whichever is longer, OR use of any investigational RSV vaccines after HCT.
2. Receiving a prescription, OTC, or herbal medication that is a potent inducer or inhibitor of CYP3A4, within 2 weeks of Randomization.
3. Receiving a prescription, OTC, or herbal medication that is a substrate of CYP3A4 with a narrow therapeutic index where monitoring blood levels is not possible.
4. Known chronic infection with hepatitis B, C, or HIV.
5. Is in the pre-engraftment period during RSV infection.
6. Admitted to the hospital primarily for lower respiratory tract disease of any cause as determined by the Investigator.
7. Any condition requiring mechanical ventilation or vasopressor support at the time of randomization.
8. Clinically significant bacteremia or fungemia within 5 days prior to Screening that has not been adequately treated.
9. Clinically significant bacterial, fungal, or viral pneumonia within 2 weeks prior to Screening that has not been adequately treated.
10. Excessive nausea/vomiting at Screening or an inability to swallow capsules.
11. Elevation of hepatic enzymes or renal compromise.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a progression to Lower Respiratory Tract Complication (LRTC) during the study | Pre-dose baseline (Day 1) through Visit 8 (Day 28)
  Progression to LRTC during the study defined as one of the following:
  * Primary LRTI caused by RSV
  * Secondary bacterial LRTI
  * LRTI caused by another pathogen
  * LRTC of unknown etiology
Change in RSV nasal viral load (via RT-qPCR) | Pre-dose baseline (Day 1) through study completion; up to Visit 8 (Day 28)
  RSV change measured by the time-weighted average (DAVG) viral load using RT qPCR

SECONDARY OUTCOMES:
Percent of participants who experience AEs, TEAEs, SAEs and withdrawals due to TEAEs | First dose of study drug through Visit 8 (Day 28)
  Safety analyses will include a summary of AEs, including but not limited to n (%) of subjects in each treatment group and overall.
Evaluate safety and tolerability of RV521 by assessing changes from baseline in systolic and diastolic BP (vital sign parameters) | Baseline through Visit 8 (Day 28)
  BP will be collected in mm Hg. Quantitative variables will be summarized used the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate safety and tolerability of RV521 by assessing changes from baseline in body temperature (vital sign parameters) | Baseline through Visit 8 (Day 28)
  Body Temperature will be collected in degrees Fahrenheit (°F) or degrees Celsius (°C). Quantitative variables will be summarized used the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate safety and tolerability of RV521 by assessing changes from baseline in respiration rate (vital sign parameters) | Baseline through Visit 8 (Day 28)
  Respiration rate will be measured in breaths per minute. Quantitative variables will be summarized used the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate safety and tolerability of RV521 by assessing changes from baseline in pulse/heart rate (vital sign parameters) | Baseline through Visit 8 (Day 28)
  Heart rate will be measured in beats per minute. Quantitative variables will be summarized used the statistics n, mean, standard deviation, median, minimum and maximum.
Evaluate safety and tolerability of RV521 by assessing changes from baseline weight/BMI | Baseline through Visit 8 (Day 28)
  Weight and height will be collected and combined to report BMI
Evaluate the proportion of subjects with changes and shifts in hematology/clinical chemistry/urinalysis laboratory values (laboratory tests read by a central lab) from baseline. | Collected at Visit 2/Day 1 (pre-dose), Visit 4/Day 3, Visit 6/Day 14 and Visit 8/Day 28
  Results at each visit will be summarized using the statistics n, mean, standard deviation, median, minimum and maximum. Also, change from baseline will also be summarized by post baseline visits.
Evaluate the proportion of subjects with changes in ECG measurements and changes in clinical impression from baseline | Measurements will be taken at Day 1/Visit 2 (pre-dose and at 5-hours post-dose), on Day 3/Visit 4 (at 5 hours post-dose), and at Visit 6 (Day 14)
  ECGs will be taken with a centrally supplied ECG machine and electronically transmitted to a central ECG repository. ECG will only be evaluated by the Investigator for normal, abnormal NCS and abnormal CS.
  Parameters collected will be:
  * Ventricular Heart Rate (bpm)
  * PR Interval (msec)
  * QRS Interval (msec)
  * QT Interval (msec)
  * QTcB Interval (msec)
  Results at each visit will be summarized using the statistics: n (number of observations), mean, SD, median, minimum and maximum.
Relationship between plasma exposures of RV521 and RSV viral loads measured in nasal swabs by RT-qPCR | Pre-dose baseline (Day 1) and every visit through Visit 8 (Day 28)
  Nasal swabs will be collected for analysis of viral load and RSV F protein gene sequencing at a central laboratory. Viral load will be assessed at intervals from nasal swabs by RT-qPCR.
Relationship between plasma exposures of RV521 and RSV viral loads measured in nasal swabs by CBIA | Pre-dose baseline (Day 1) and every visit through Visit 8 (Day 28)
  Nasal swabs will be collected for analysis of viral load and RSV F protein gene sequencing at a central laboratory. Viral load will be assessed at intervals from nasal swabs by CBIA.
Mean change in RSV viral load assessed via CBIA | Pre-dose baseline (Day 1) through study completion; up to Visit 8 (Day 28)
  change measured by the time weighted average (DAVG) viral load using CBIA
Mean change from baseline in viral RNA shedding | Pre-dose baseline (Day 1) through study completion; up to Visit 8 (Day 28)
  RSV assessed via nasal swabs collected at each visit and analyzed at a central laboratory.
Proportion of subjects who no longer shed RSV assessed by both RT-qPCR and CBIA at each timepoint | Pre-dose baseline (Day 1) through study completion; up to Visit 8 (Day 28)
  RSV assessed via nasal swabs collected at each visit and analyzed at a central laboratory.
Time to improvement in RSV-related symptoms | Daily from baseline (Day 1) through Visit 8 (Day 28)
  Defined as all symptoms present at initiation of therapy are mild or no longer present. (absent/resolved)
Time to total resolution of all RSV-related symptoms | Daily from baseline (Day 1) through Visit 8 (Day 28)
  Defined as all symptoms are no longer present.
Proportion of days with lowest daily SpO2 ≥ 90% on room air | Daily from baseline (Day 1) through Visit 8 (Day 28)
  SpO2 measured at every visit. For subjects on oxygen or who are mechanically ventilated may have this waived.
Number of days where supplementary oxygen was required | Baseline (Day 1) through Visit 8 (Day 28)
  Use of daily supplementary oxygen will be collected throughout the study.
Proportion of subjects who require hospitalization during the study | Baseline (Day 1) through Visit 8 (Day 28)
  Daily hospitalization utilization will be collected
Mean number of days of hospitalization during the study | Baseline (Day 1) through Visit 8 (Day 28)
  Daily hospitalization utilization will be collected
Proportion of subjects requiring ICU | Baseline (Day 1) through Visit 8 (Day 28)
  Daily ICU utilization will be collected
Mean number of days in ICU | Baseline (Day 1) through Visit 8 (Day 28)
  Daily ICU utilization will be collected
Proportion of subjects requiring mechanical ventilation | Baseline (Day 1) through Visit 8 (Day 28)
  Daily mechanical ventilation requirements will be collected
Number of subjects who experience death (all-cause mortality) | First dose of study drug through Visit 8 (Day 28)
  Patient outcome will be followed and collected
Number of subjects who experience death attributable to LRTC | First dose of study drug through Visit 8 (Day 28)
  Patient outcome will be followed and collected

CONTACTS AND LOCATIONS:
Overall Officials: PfizerCT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests